CLINICAL TRIAL: NCT06719375
Title: Evaluation of Gait Impairment and Correlation With Clinical Assessment Tools Before and After Surgery in Patients With Cervical Myelopathy Using Inertial Sensors
Brief Title: Evaluation of Gait Impairment and Correlation in Patients With DCM
Acronym: DCM-HFIMU
Status: Not yet recruiting | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sungchul Huh, Assistant Professor, Department of Rehabilitation Medicine, Pusan National University Yangsan Hospital
Other Study IDs: 2024-0053
Record Dates: First submitted 2024-11-28; First posted 2024-12-05 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Myelopathy Cervical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 50 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Degenerative Cervical Myelopathy (DCM) Patients: Patients diagnosed with Degenerative Cervical Myelopathy (DCM) scheduled for surgery. This group will undergo gait analysis and clinical assessments at three time points: 10 days pre-surgery, 10 days post-surgery, and 30 days post-surgery.
  Interventions: Device: Gait Analysis Using IMU Sensor

INTERVENTIONS:
Device: Gait Analysis Using IMU Sensor — Inertial Measurement Unit (IMU) sensor-based 3D gait analysis to assess spasticity and gait impairment. This intervention aims to provide quantitative data on gait parameters in DCM patients before and after surgery.

SUMMARY:
This study aims to evaluate gait impairment in patients with Degenerative Cervical Myelopathy (DCM) before and after surgery using an inertial measurement unit (IMU) sensor. By comparing IMU-derived gait parameters with traditional clinical assessment tools (e.g., Modified Ashworth Scale, mJOA, and GRASSP), the study seeks to determine the effectiveness and reliability of IMU sensors for assessing and monitoring gait improvement and neurological recovery in DCM patients. This study is conducted outside the United States and does not involve interventions or devices subject to U.S. FDA regulation.

DETAILED DESCRIPTION:
This observational study will investigate the correlation between gait parameters measured with an IMU sensor and established clinical evaluation tools for patients with Degenerative Cervical Myelopathy (DCM). The primary aim is to quantify gait impairments before and after surgical intervention and to verify the IMU sensor's utility as a quantitative assessment tool. The study will recruit both DCM patients and a control group to evaluate the sensitivity of the IMU sensor in detecting fine motor and gait differences. Outcomes will be analyzed using statistical comparisons of pre- and post-surgery measurements, with specific focus on gait speed, cadence, stride length, and spasticity. The anticipated goal is to validate the IMU sensor as a reliable alternative to existing clinical tools, facilitating early detection of gait impairment and monitoring post-surgical improvement in DCM patients. This study is conducted entirely outside the United States and does not involve interventions or devices subject to U.S. FDA regulation. The devices and procedures used in this study are approved by local regulatory authorities in the country where the study is conducted. The study complies with applicable international and local guidelines rather than U.S. FDA requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Able to communicate and provide informed consent.
* Capable of walking at least 3 meters without assistance from others or walking aids.
* No prior surgical treatment for cervical myelopathy.
* Lower limb motor function score of 2 or higher on the mJOA scale.

Exclusion Criteria:

* Presence of severe respiratory or cardiac conditions that impede safe walking.
* Musculoskeletal issues, such as spinal deformities, affecting gait.
* History of neurological disorders affecting gait, including peripheral nerve injury, joint stiffness, stroke, traumatic brain injury, myelitis, or Parkinson's disease.
* Prior orthopedic or neurosurgical interventions that could impact gait.
* Cervical conditions resulting from trauma (acute fracture or acute disc herniation), tumor, or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults aged 18 years or older who are diagnosed with cervical myelopathy and exhibit gait disturbances. Participants must be capable of walking at least 3 meters unassisted and have not undergone previous surgical treatment for cervical myelopathy. This population will be assessed using gait analysis and clinical evaluation tools to measure gait parameters and motor function. Individuals with severe respiratory or cardiac conditions, musculoskeletal issues affecting gait, or a history of neurological disorders impacting mobility will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Step Length | 10 days before surgery, 10 days after surgery, and 30 days after surgery.
  Step length is measured in centimeters (cm) to independently evaluate the gait characteristics of patients with Degenerative Cervical Myelopathy (DCM). Step length is defined as the distance covered between two successive placements of the same foot and is a critical parameter to assess balance and mobility.
Walking Speed | 10 days before surgery, 10 days after surgery, and 30 days after surgery.
  Walking speed is measured in kilometers per hour (km/h) to independently assess the gait characteristics of patients with Degenerative Cervical Myelopathy (DCM). Walking speed evaluates the efficiency of ambulation over a defined distance and is a vital measure of functional mobility.
Stride Length | 10 days before surgery, 10 days after surgery, and 30 days after surgery.
  Stride length is measured in centimeters (cm) to independently evaluate the gait characteristics of patients with Degenerative Cervical Myelopathy (DCM). Stride length is defined as the distance covered in one complete gait cycle and provides insights into the patient's walking stability.
Cadence | 10 days before surgery, 10 days after surgery, and 30 days after surgery.
  Cadence is measured in steps per minute (steps/min) to independently assess the gait characteristics of patients with Degenerative Cervical Myelopathy (DCM). Cadence represents the number of steps taken per minute and is used to analyze walking rhythm and patterns.

SECONDARY OUTCOMES:
Modified Japanese Orthopaedic Association (mJOA) Score | 10 days before surgery, 10 days after surgery, and 30 days after surgery.
  The mJOA score is used to assess neurological function in patients with Degenerative Cervical Myelopathy (DCM). This score evaluates motor dysfunction, sensory dysfunction, and bladder function. The score ranges from 0 (worst outcome) to 18 (best outcome), with higher scores indicating better neurological function.
Modified Ashworth Scale (MAS) | 10 days before surgery, 10 days after surgery, and 30 days after surgery.
  The MAS score is used to assess spasticity in patients with Degenerative Cervical Myelopathy (DCM). The scale ranges from 0 (no increase in muscle tone) to 4 (rigid in flexion or extension). Lower scores indicate better outcomes, reflecting reduced spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Sungchul Huh, PhD, Principal Investigator — Pusan National University Yangsan Hospital

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared to protect the privacy and confidentiality of participants. Due to the sensitive nature of the medical data involved, and to comply with institutional policies and ethical standards, data sharing is restricted to ensure the security and anonymity of participant information.

REFERENCES:
- [Background] Moorthy RK, Bhattacharji S, Thayumanasamy G, Rajshekhar V. Quantitative changes in gait parameters after central corpectomy for cervical spondylotic myelopathy. J Neurosurg Spine. 2005 Apr;2(4):418-24. doi: 10.3171/spi.2005.2.4.0418. PMID 15871480
- [Background] Lee DH, Yoo JY, Cho JH, Hwang CJ, Lee CS, Kim C, Ha JK, Park KB. Subclinical gait disturbance and postoperative gait improvement in patients with degenerative cervical myelopathy. Sci Rep. 2021 May 27;11(1):11179. doi: 10.1038/s41598-021-90884-2. PMID 34045643
- [Background] Maezawa Y, Uchida K, Baba H. Gait analysis of spastic walking in patients with cervical compressive myelopathy. J Orthop Sci. 2001;6(5):378-84. doi: 10.1007/s007760170002. PMID 11845345
- [Background] Siasios ID, Spanos SL, Kanellopoulos AK, Fotiadou A, Pollina J, Schneider D, Becker A, Dimopoulos VG, Fountas KN. The Role of Gait Analysis in the Evaluation of Patients with Cervical Myelopathy: A Literature Review Study. World Neurosurg. 2017 May;101:275-282. doi: 10.1016/j.wneu.2017.01.122. Epub 2017 Feb 9. PMID 28192261
- [Background] Malone A, Meldrum D, Bolger C. Three-dimensional gait analysis outcomes at 1 year following decompressive surgery for cervical spondylotic myelopathy. Eur Spine J. 2015 Jan;24(1):48-56. doi: 10.1007/s00586-014-3267-1. Epub 2014 Mar 13. PMID 24622959
- [Background] Williams G, Morris ME, Schache A, McCrory P. Observational gait analysis in traumatic brain injury: accuracy of clinical judgment. Gait Posture. 2009 Apr;29(3):454-9. doi: 10.1016/j.gaitpost.2008.11.005. Epub 2008 Dec 23. PMID 19109020
- [Background] McGinley JL, Baker R, Wolfe R, Morris ME. The reliability of three-dimensional kinematic gait measurements: a systematic review. Gait Posture. 2009 Apr;29(3):360-9. doi: 10.1016/j.gaitpost.2008.09.003. Epub 2008 Nov 13. PMID 19013070
- [Background] Malone A, Meldrum D, Bolger C. Gait impairment in cervical spondylotic myelopathy: comparison with age- and gender-matched healthy controls. Eur Spine J. 2012 Dec;21(12):2456-66. doi: 10.1007/s00586-012-2433-6. Epub 2012 Jul 24. PMID 22825630
- [Background] Mandelli F, Zhang Y, Nuesch C, Ewald H, Aghlmandi S, Halbeisen F, Scharen S, Mundermann A, Netzer C. Gait function assessed using 3D gait analysis in patients with cervical spinal myelopathy before and after surgical decompression: a systematic review and meta-analysis. Spine J. 2024 Mar;24(3):406-416. doi: 10.1016/j.spinee.2023.09.030. Epub 2023 Oct 21. PMID 37866484